CLINICAL TRIAL: NCT05140733
Title: Cost-effectiveness Analysis Between Lumbar Foraminotomy and Lumbar Single or Double Levels Fusion Surgery in Patients With Foraminal Stenosis
Brief Title: Outcomes of Patients With Foraminal Stenosis
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chi Heon Kim, Professor, Seoul National University Hospital
Other Study IDs: Foraminotomy
Record Dates: First submitted 2021-08-22; First posted 2021-12-01 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Foraminal Stenosis
Keywords: Cost-effectiveness; surgery; deformity
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fusion: 1 or 2 levels fusion surgery
  Interventions: Procedure: Fusion surgery
- Foraminotomy: 1 or 2 levels lumbar foraminotomy
  Interventions: Procedure: lumbar foraminal decompression

INTERVENTIONS:
Procedure: lumbar foraminal decompression — lumbar foraminal decompression with endoscopic instruments.
  Groups: Foraminotomy
Procedure: Fusion surgery — Fusion surgery for patients with foraminal stenosis
  Groups: Fusion

SUMMARY:
The present study was to see the effect of minimally invasive neural foraminotomy for lumbar foraminal stenosis with unilateral radicular pain. Traditionally, fusion was was done for the patients, but recent development enable surgeon to decompress neural foramen without rigid spinal fusion. Although, clinical effect of neural foraminotomy may have limitation in attaining a comparable result to fusion surgery, a cost-effective analysis may reveal a result in a different perspective. In this regard, we designed a prospective cohort study to see the cost-effectiveness of neural foraminotomy compared to fusion surgery.

DETAILED DESCRIPTION:
Control: 1-2 levels fusion surgery Intervention: neural foraminotomy

Inclusion patients between 40 - 100 years. No improvement despite nonsurgical treatment for more than 3 months. No history of lumbar fusion surgery Single or double-level lumbar foraminal stenosis with corresponding leg pain

Exclusion Severe neurological deficit (motor grade less than Grade III) Combined inflammatory joint disease Combined neurodegenerative disease such as Parkinson's disease or dementia Combined cancer, traumatic fracture marked spinal deformity (C7 sagittal vertical axis > 10cm)

Surgery and follow-up Patients underwent foraminotomy and visits outpatient clinical at determined time points (postoperative month 1, 6, 12 and 24 months) Their clinical outcomes were recorded at each visit. Their medical costs were retrieved at the time of analysis by using hospital records.

Statistical analysis means: T-test

ELIGIBILITY:
Inclusion:

* patients between 40 - 100 years.
* No improvement despite nonsurgical treatment for more than 3 months.
* No history of lumbar fusion surgery.
* Single or double-level lumbar foraminal stenosis with corresponding leg pain

Exclusion:

* Severe neurological deficit (motor grade less than Grade III)
* Combined inflammatory joint disease
* Combined neurodegenerative disease such as Parkinson's disease or dementia * Combined cancer, traumatic fracture
* Marked spinal deformity (C7 sagittal vertical axis > 10cm)

Ages: 40 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 26 patients in each foraminotomy and fusion group.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-08-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness | preoperation
  cost to increased one quality adjusted life year (QALY) after surgical treatment
Cost-effectiveness | postoperative 6 months
  cost to increased one quality adjusted life year (QALY) after surgical treatment
Cost-effectiveness | postoperative 1 year
  cost to increased one quality adjusted life year (QALY) after surgical treatment
Cost-effectiveness | postoperative 2 years
  cost to increased one quality adjusted life year (QALY) after surgical treatment

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | preoperation
  ODI was recorded at preoperation, postoperative 6 months, 1 year and 2 years.
Oswestry disability index (ODI) | postoperative 6 months
  ODI was recorded at preoperation, postoperative 6 months, 1 year and 2 years.
Oswestry disability index (ODI) | postoperative 1 year
  ODI was recorded at preoperation, postoperative 6 months, 1 year and 2 years.
Oswestry disability index (ODI) | postoperative 2 years
  ODI was recorded at preoperation, postoperative 6 months, 1 year and 2 years.
Numeric rating scale(NRS) of pain on back (NRS-B) and legs (NRS-L) | preoperation
  NRS-B and NRS-L were recorded at preoperation, postoperative 6 months, 1 year and 2 years.
  Numeric rating scale (NRS)
  : Scale from 0 to 10. Zero means there's no pain and 10 means the maximum pain.
Numeric rating scale(NRS) of pain on back (NRS-B) and legs (NRS-L) | postoperative 6 months
  NRS-B and NRS-L were recorded at preoperation, postoperative 6 months, 1 year and 2 years.
  Numeric rating scale (NRS)
  : Scale from 0 to 10. Zero means there's no pain and 10 means the maximum pain.
Numeric rating scale(NRS) of pain on back (NRS-B) and legs (NRS-L) | postoperative 1 year
  NRS-B and NRS-L were recorded at preoperation, postoperative 6 months, 1 year and 2 years.
  Numeric rating scale (NRS)
  : Scale from 0 to 10. Zero means there's no pain and 10 means the maximum pain.
Numeric rating scale(NRS) of pain on back (NRS-B) and legs (NRS-L) | postoperative 2 years.
  NRS-B and NRS-L were recorded at preoperation, postoperative 6 months, 1 year and 2 years.
  Numeric rating scale (NRS)
  : Scale from 0 to 10. Zero means there's no pain and 10 means the maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes
I am willing to share all data after publication.
Supporting Information: Study Protocol, SAP
Time Frame: after publication of study results.